CLINICAL TRIAL: NCT02544165
Title: Non Invasive Measurement of the Haemodynamic Parameters and of the Advanced Glycation End Products (AGEs) Levels in Students Smokers and in Students Who Intake Caffeine (NONINVASHAEMOAGES)
Brief Title: Non Invasive Measurement of the Haemodynamic Parameters and of the Advanced Glycation End Products (AGEs) Levels
Acronym: NONINVASHEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Education Institute of Sterea Ellada (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, ANNA DELTSIDOU, Associate Professor, Technological Education Institute of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0925-0586
Record Dates: First submitted 2015-08-22; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Hemodynamic Instability; Skin and Subcutaneous Tissue Disorders
Keywords: smoking; caffeine intake; haemodynamic parameters; Advanced Glycation End Products (AGEs); Non-invasive measurements devices
MeSH Terms: conditions — Skin Diseases; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Caffeine intake (Experimental): 100mg of Caffeine intake
  Interventions: Dietary Supplement: caffeine intake
- Cigarette smoking (Experimental): smoking of one cigarette
  Interventions: Other: cigarette smoking
- Caffeine intake and Cigarette smoking (Experimental): 100mg of Caffeine intake and smoking of one cigarette
  Interventions: Other: cigarette smoking; Other: Caffeine intake and Cigarette smoking
- Control group (No Intervention): no intervention group

INTERVENTIONS:
Dietary Supplement: caffeine intake — The subjects of this group should intake 100 mg of caffeine after the first measurement of haemodynamic parameters with the Finometer device and after the first measurement of the advanced glycation end products accumulation with AgeReader device.
  Arms: Caffeine intake
Other: cigarette smoking — The subjects of this group should smoke one cigarette after the first measurement of haemodynamic parameters with the Finometer device and after the first measurement of the advanced glycation end products accumulation with AgeReader device.
  Arms: Caffeine intake and Cigarette smoking; Cigarette smoking
Other: Caffeine intake and Cigarette smoking — The subjects of this group should smoke one cigarette and should consume 100 mg of caffeine after the first measurement of haemodynamic parameters with the Finometer device and after the first measurement of the advanced glycation end products accumulation with AgeReader device.
  Arms: Caffeine intake and Cigarette smoking

SUMMARY:
The aim of this study was to investigate the difference in accumulation of AGEs (advanced glycation end-products) in the tissues of individuals who smoke in comparison with individuals who do not as well as of individuals who consume caffeine versus those who do not, and finally to examine the probable differences concerning participants' haemodynamic parameters.

DETAILED DESCRIPTION:
Materials and methods Study population The study population consisted of students of Health Care Professions who accepted to participate in the study and gave their informed consent for their participation. The population study included healthy volunteers without cardiovascular problems, other chronic or systemic diseases. Participants were divided into 3 intervention groups: the first group are non-smokers who consume caffeine on daily basis, the second group are smokers who do not consume caffeine on daily basis, and the third group are smokers who consume caffeine on daily basis. Additionally, there was a control group consisting of non smoking students and no caffeine users on daily basis.

Methodology A complete medical history with information about the health status of the subjects, drug use and the main risk factors for cardiovascular conditions was recorded. Details concerning smoking and drinking habits, caffeine intake and other medical conditions and conditions from the individual and family history were retrieved, by filling-in self-reporting questionnaires. Information about dietary habits and physical activity of the subjects was also recorded. Body weight and height of all participants were measured. Also, participants were informed that on the day of the scheduled measurements, they should not have breakfast nor smoke for 2 hours (for smokers) prior to measurements and finally abstain from any physical activity. Inclusion criteria in the group of smokers were cigarette smoking of more than 10 cigarettes/day for at least 2 years.

Skin- autofluorescence measurement Tissue AGEs accumulation was assessed using a validated skin-autofluorescence (skin-AF) device, namely AGE Reader. In short, the AGE reader illuminates a skin surface of approximately 4 cm2, guarded against surrounding light, with an excitation light source between 300 and 420 nm (peak excitation ~370 nm). Skin-AF was measured at the volar side of the lower arm at approximately 10-15 cm below the elbow fold. Care had been taken to perform the measurement at normal skin site (without visible vessels, scars, lichenification, or other skin abnormalities). The investigators performed three measurements with a 5min interval between them and the investigators calculated the mean value of three measurements. For the individuals who smoked, these measurements were repeated 2 hours after the smoking of one cigarette and for individuals who consumed caffeine, measurements were repeated after the intake of 100 mg caffeine (delivered as a beverage). This was done to check whether there was a change in accumulation of AGEs following cigarette smoking and caffeine intake.

Haemodynamic parameters' measurement The haemodynamic parameters' measurement included measurement of cardiac output, stroke volume, systolic and diastolic blood pressure, mean pressure, pulse rate, interbeat intervals, arterial compliance and systemic vascular resistance. These measurements were performed with the Finometer device (FMS, Finapress Medical System, BV, Netherlands), while the data were recorded by using the Beatscope, a specially designed software, to transfer data to the PC and to process pressure waveform files. The measurements were performed by using a non-invasive method via a finger cuff, which was wrapped around the finger of the individual, who was in a lying down position for 10 min before the measurements in a room of a sound-attenuated, temperature-controlled environment, in order to ensure that all measurements will be performed under constant and stable conditions. Subsequently, the haemodynamic parameters' measurement was performed for 15 min in a sitting position. Additionally, for smokers the measurements were repeated after 15-30 min since smoking one cigarette and after 45 min for individuals who consumed caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals who smoke ≥ 10 cigarettes per day
* Healthy non smoking individuals consuming caffeine on daily basis
* Healthy individuals, smoking and consuming caffeine on daily basis

Exclusion Criteria:

* Individuals suffering from any chronic disease (diabetes mellitus, cardiovascular diseases, etc)

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Measurements of the haemodynamic parameters and accumulation of AGEs before smoking and before intake of caffeine | 0 min
  Measurements of the haemodynamic parameters and accumulation of AGEs before smoking of one cigarette and consumption of 100 mg caffeine

SECONDARY OUTCOMES:
Changes in the haemodynamic parameters and accumulation of AGEs after consuming 100 mg of caffeine | 60 min
  Measurement of haemodynamic parameters with finometer device in 45 min after consuming of 100 mg caffeine and measurement of the accumulation of AGEs with the device AgeReader
Changes in the haemodynamic parameters and accumulation of AGEs after smoking of one cigarette | 60 min
  Measurement of haemodynamic parameters with finometer device in 45 min after the smoking of one cigarette and measurement of the accumulation of AGEs with the device AgeReader
Changes in the haemodynamic parameters and in the accumulation of AGEs after smoking of one cigarette and after consuming of 100 mg caffeine | 60 min
  Measurement of haemodynamic parameters with finometer device in 45 min after the smoking of one cigarette and measurement of the accumulation of AGEs with the device AgeReader

CONTACTS AND LOCATIONS:
Overall Officials: Anna Deltsidou, PhD, Study Director — Technological Educational Institute of Athens, Greece
Locations (1):
- Technological Educational Institute of Sterea Ellada, Lamia, Greece